CLINICAL TRIAL: NCT04762433
Title: Parallel-Group, Randomised Single-centred, Single-blind, Pilot and Feasibility Study for KEPT-app Trial: Study Protocol
Brief Title: Kegel Exercise Pregnant Training mHealth App
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Aida Jaffar, Investigator and Family Medicine Specialist, PhD Doctorate, Psuchiatry Department, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NMRR-19-471-45606
Record Dates: First submitted 2021-02-09; First posted 2021-02-21 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Pregnancy Related; Urinary Incontinence
Keywords: Pilot study; Feasibility study; Acceptability; mHealth app; Pelvic Floor Muscle Training
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Intervention Model Description: This study will use a single-blind, single-centre, parallel, randomized controlled trial (RCT) design which will incorporate individualised treatment flexibility, as in a real-world setting, and provide a realistic estimation in future KEPT-app RCT study (Sidik et al., 2021).
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigator and the assessor will be blinded as to the recruitment and allocation via the electronic consent format and the intervention via the mobile application.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kegel Exercise Pregnancy Training - App (Experimental): The intervention arm will be given a mHealth app for two months duration with the usual antenatal follow-up.
  Interventions: Device: Kegel Exercise Pregnancy Training - app
- Waitlist control (No Intervention): The control (waitlist) group will continue their usual antenatal follow-up and the KEPT-app will be given after the study ends.

INTERVENTIONS:
Device: Kegel Exercise Pregnancy Training - app — KEPT-app is designed to educate pregnant women on PFMT via the step-by-step training with the capability element to improve their confidence and skills (beginner, intermediate and advance skills). Pregnant women are encouraged to continue adopt the PFMT throughout pregnancy until postpartum period.
  The details of the mHealth app content was developed based on the need assessment gathered from the cross-sectional study (Jaffar et al., 2020). It was conducted to identify the need of PFMT by looking at the prevalence of the UI among pregnant women and to understand their knowledge, attitude, and practices towards PFMT.
  Arms: Kegel Exercise Pregnancy Training - App

SUMMARY:
This pilot feasibility study protocol is to assess the feasibility in the future definitive trial that is the Kegel Exercise Pregnancy Training app (KEPT-app) trial. The aim of this study as follows: (1) to evaluate the recruitment capability of the pregnant women, (2) to evaluate the acceptability of the KEPT-app, (3) to determine the implementation feasibility of using KEPT-app, and (4) to determine the preliminary effectiveness of KEPT-app to improve PFMT skills of pregnant women.

DETAILED DESCRIPTION:
The aim of this pilot feasibility study as follows: (1) to evaluate the recruitment capability of the pregnant women, (2) to evaluate the acceptability of the KEPT-app, (3) to determine the implementation feasibility of using KEPT-app, and (4) to determine the preliminary effectiveness of KEPT-app to improve PFMT skills of pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women at 26-27 weeks of gestation, any parity with either stress UI or mixed UI will be included.
* Participants are Malaysian citizens who consist of Malay, Chinese, Indian, and native ethnicities.

Exclusion Criteria:

* pregnant women with a chronic medical problem(s) before pregnancy, complicated pregnancies or conditions which are not advisable to practise PFMT will be excluded.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 26 (Actual)
Dates: Start 2021-05-17 (Actual); Primary Completion 2021-11-17 (Actual); Study Completion 2021-11-17 (Actual)

PRIMARY OUTCOMES:
Acceptability of the mHealth app intervention. | 2 months
  Interactive Malay-mHealth App Usability Questionnaire Standardized outcome measure with additional Qualitative data collection
  1. How many stars would you recommend this app to your friends?
  2. How many stars would you rate the content of this app?
  3. How many stars would you rate the comfort of using this app?
  4. How many stars would you rate simplicity using this app?
  5. How many stars would you rate the recruitment process using this app?
  6. How many stars would you rate the quality of the app?
  7. Factors influenced/hindered using this app?
  8. What motivates you to continue the PFMT? (Further information will be collected via qualitative data feedback)

SECONDARY OUTCOMES:
Validation of educational video | 1 month
  Patient Educational Material Assessment Tool (PEMAT) Standardized outcome measure
Kegel's exercise adherence | 1 month and 2 months
  Exercise Adherence Rating Scale Standardized outcome measure where the increasing PFMT adherence from lowest score (0) to maximum score (24) of Exercise Adherence Rating Scale (EARS) Increasing Exercise adherence from lowest score (0) to maximum score (24).
Self-efficacy towards Kegel's Exercise | 1 month and 2 months
  Self-Efficacy Scale For Practicing Pelvic Floor Exercise Questionnaire Standardized outcome measure The final scores were obtained by calculating the mean of the items, ranging between 0 and 100, in which the higher values were equivalent to higher self-efficacy in practising PFME.
Urinary incontinence | 1 month and 2 months
  International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-UI SF) The overall score is between 0 and 21 whereby greater values of the overall scores indicated increased severity of UI.
Knowledge, Attitude and Practice Pelvic Floor Muscle Training | 1 month and 2 months
  The overall knowledge scores ranged between 0 and 14, and a higher score suggested a higher level of knowledge. The total scores for attitude ranged between 8 and 40, with higher scores suggesting a positive attitude. The total scores for the practice domain ranged between 4 and 16, and the higher score suggested higher levels of its practice.
Quality of Life of pregnant women | 1 month and 2 months
  The minimum mark was 19 and the maximum mark was 76 indicating severely affecting QOL using the Incontinence Impact Questionnaire Quality of Life (ICIQ-LUTSqol).

CONTACTS AND LOCATIONS:
Overall Officials: Sherina Mohd Sidik, PhD, Principal Investigator — Universiti Putra Malaysia
Locations (1):
- (Health Clinic Ampang) Ministry of Health, Hulu Langat, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No
The data will be collected via the KEPT-app link entered directly into the trial database. Data gathered from the KEPT-app enables the participants to access their data, monitor their UI symptoms and act as PFMT motivation. The data will be stored in the cloud-based Azure storage.

REFERENCES:
- [Background] Sidik SM, Jaffar A, Foo CN, Muhammad NA, Abdul Manaf R, Ismail SIF, Alagirisamy P, Ahmad Fazlah AF, Suli Z, Goodyear-Smith F. KEPT-app trial: a pragmatic, single-blind, parallel, cluster-randomised effectiveness study of pelvic floor muscle training among incontinent pregnant women: study protocol. BMJ Open. 2021 Jan 12;11(1):e039076. doi: 10.1136/bmjopen-2020-039076. PMID 33436465
- [Background] Mustafa N, Safii NS, Jaffar A, Sani NS, Mohamad MI, Abd Rahman AH, Mohd Sidik S. Malay Version of the mHealth App Usability Questionnaire (M-MAUQ): Translation, Adaptation, and Validation Study. JMIR Mhealth Uhealth. 2021 Feb 4;9(2):e24457. doi: 10.2196/24457. PMID 33538704
- [Background] Jaffar A, Mohd Sidik S, Foo CN, Muhammad NA, Abdul Manaf R, Fadhilah Ismail SI, Suhaili N. Protocol of a Single-Blind Two-Arm (Waitlist Control) Parallel-Group Randomised Controlled Pilot Feasibility Study for mHealth App among Incontinent Pregnant Women. Int J Environ Res Public Health. 2021 Apr 30;18(9):4792. doi: 10.3390/ijerph18094792. PMID 33946203
- [Background] Jaffar A, Mohd-Sidik S, Foo CN, Admodisastro N, Abdul Salam SN, Ismail ND. Improving Pelvic Floor Muscle Training Adherence Among Pregnant Women: Validation Study. JMIR Hum Factors. 2022 Feb 3;9(1):e30989. doi: 10.2196/30989. PMID 35113025
- [Background] Jaffar A, Mohd-Sidik S, Abd Manaf R, Foo CN, Gan QF, Saad H. Quality of life among pregnant women with urinary incontinence: A cross-sectional study in a Malaysian primary care clinic. PLoS One. 2021 Apr 28;16(4):e0250714. doi: 10.1371/journal.pone.0250714. eCollection 2021. PMID 33909678
- [Background] Jaffar A, Mohd-Sidik S, Nien FC, Fu GQ, Talib NH. Urinary incontinence and its association with pelvic floor muscle exercise among pregnant women attending a primary care clinic in Selangor, Malaysia. PLoS One. 2020 Jul 15;15(7):e0236140. doi: 10.1371/journal.pone.0236140. eCollection 2020. PMID 32667936
- [Background] Jaffar, A., Mohd Sidik, S., Admodisastro, N., Mansor, E. I., & Chia Fong, L. Expert's Usability Evaluation of the Pelvic Floor Muscle Training mHealth App for Pregnant Women. International Journal of Advanced Computer Science and Applications. 2021; 12(10), 165-173.
- [Background] Sacomori C, Cardoso FL, Porto IP, Negri NB. The development and psychometric evaluation of a self-efficacy scale for practicing pelvic floor exercises. Braz J Phys Ther. 2013 Jul-Aug;17(4):336-42. doi: 10.1590/S1413-35552013005000104. Epub 2013 Aug 30. English, Portuguese. PMID 24072223
- [Background] Sacomori C, Berghmans B, Mesters I, de Bie R, Cardoso FL. Strategies to enhance self-efficacy and adherence to home-based pelvic floor muscle exercises did not improve adherence in women with urinary incontinence: a randomised trial. J Physiother. 2015 Oct;61(4):190-8. doi: 10.1016/j.jphys.2015.08.005. Epub 2015 Sep 11. PMID 26365268
- [Background] Asklund I, Nystrom E, Sjostrom M, Umefjord G, Stenlund H, Samuelsson E. Mobile app for treatment of stress urinary incontinence: A randomized controlled trial. Neurourol Urodyn. 2017 Jun;36(5):1369-1376. doi: 10.1002/nau.23116. Epub 2016 Sep 9. PMID 27611958
- [Background] Lim R, Liong ML, Lau YK, Yuen KH. Validity, reliability, and responsiveness of the ICIQ-UI SF and ICIQ-LUTSqol in the Malaysian population. Neurourol Urodyn. 2017 Feb;36(2):438-442. doi: 10.1002/nau.22950. Epub 2015 Dec 23. PMID 26693962
- [Background] Julious, S. A. Sample size of 12 per group rule of thumb for a pilot study. Pharmaceutical Statistics: The Journal of Applied Statistics in the Pharmaceutical Industry. 2005; 4(4), 287-291.
- [Background] Jaffar A, Tan CE, Mohd-Sidik S, Admodisastro N, Goodyear-Smith F. Persuasive Technology in an mHealth App Designed for Pelvic Floor Muscle Training Among Women: Systematic Review. JMIR Mhealth Uhealth. 2022 Mar 22;10(3):e28751. doi: 10.2196/28751. PMID 35315777
- [Result] Jaffar A, Mohd Sidik S, Foo CN, Muhammad NA, Abdul Manaf R, Suhaili N. Preliminary Effectiveness of mHealth App-Based Pelvic Floor Muscle Training among Pregnant Women to Improve Their Exercise Adherence: A Pilot Randomised Control Trial. Int J Environ Res Public Health. 2022 Feb 18;19(4):2332. doi: 10.3390/ijerph19042332. PMID 35206520
- [Result] Jaffar A, Muhammad NA, Mohd Sidik S, Admodisastro N, Abdul Manaf R, Foo CN, Suhaili N. Feasibility and Usability of Kegel Exercise Pregnancy Training App (KEPT App) among Pregnant Women with Urinary Incontinence. Int J Environ Res Public Health. 2022 Mar 17;19(6):3574. doi: 10.3390/ijerph19063574. PMID 35329262